CLINICAL TRIAL: NCT01921036
Title: Individuell Dosiertes Kraft-ausdauer-training in Ambulanten Herzgruppen - Einfluss Auf Koerperliche Belastbarkeit Von Herzpatienten.
Brief Title: The Effects of Combined Exercise Training on Exercise Capacity in Cardiac Rehabilitation
Acronym: DOPPELHERZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2931/10; DRKS00003625 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2013-07-05; First posted 2013-08-13 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combined exercise (Experimental): 90 minutes combined endurance and resistance exercise once a week plus 90 minutes traditional cardiac rehabilitation once a week over six months
  Interventions: Procedure: combined exercise
- traditional cardiac rehabilitation (Active Comparator): The group-based program is offered for 90 minutes twice a week and is a combination of gymnastics, coordination and flexibility exercises, and includes educational components targeting diet and nutrition, stress and relaxation, methods for coping with CVD and behavioral and lifestyle change.
  Interventions: Procedure: traditional cardiac rehabilitation

INTERVENTIONS:
Procedure: traditional cardiac rehabilitation — mutifactoral cardiac rehabilitation
  Arms: traditional cardiac rehabilitation
Procedure: combined exercise — Moderate endurance and resistance exercise once a week over six months
  Arms: combined exercise

SUMMARY:
Seventy patients in cardiac rehabilitation with maximal exercise capacity less than 1.4 watt per kilogram bodyweight will be randomized 1:1 into either an intervention training (IN) group or usual care (UC). The IN patients will perform supervised endurance and resistance exercise for approximately 90 minutes once a week and traditional cardiac rehabilitation (TCR) once a week; the UC patients will perform TCR twice a week. The intervention is planned for six months with a follow-up of a further six months. The primary investigation is differences between IN and UC with regard to changes in exercise capacity (max watt/kgBW).

DETAILED DESCRIPTION:
The DOPPELHERZ (The influence of individualized resistance-endurance exercise training on maximal power output in outpatient cardiac rehabilitation) randomized controlled trial was performed at the Department of Prevention and Sports Medicine, Klinikum rechts der Isar in Munich, Germany. 70 patients eligible for and/or participating in cardiac rehabilitation were randomized to six months in an individualized combined exercise group (ICE) or group- based cardiac rehabilitation (GCR), considered usual care in this patient population.

All patients gave written informed consent, the study protocol was approved by the local university hospital ethics committee, all procedures were conducted according to the Declaration of Helsinki.

Participants: All patients were American Heart Association Class "C" (moderate to high risk) based on the presence of cardiac disease and maximal power output of <5 METs (corresponding to <1.4 W/kg body weight), who met eligibility criteria for CR at the time of recruitment. Patients with decompensated or highly symptomatic (NYHA IV) heart failure, acute illness or injury, cardiac hospitalizations within six weeks of inclusion, drug abuse, unstable blood pressure or arrhythmias, high grade valve stenosis or instable diabetes mellitus were excluded.

Primary endpoint: The primary endpoint was change in maximal relative power output (W/kg) measured by CPX after six months.

Exercise training program In both the intervention and usual care arms of the study, exercise training was prescribed twice weekly over a period of six months, and all exercise sessions were led by certified exercise instructors and monitored by physicians.

Group-based cardiac rehabilitation (GCR): The GCR group performed regular exercise in a state-sanctioned cardiac rehabilitation group. This form of GCR is considered Phase III aftercare and has been described elsewhere9. Briefly, GCR patients received moderate-intensity heart rate targets from exercise cardiologists based on CPX results. The group-based program is offered for 90 minutes twice a week and is a combination of gymnastics (including endurance and resistance components), coordination and flexibility exercises, and includes educational components targeting diet and nutrition, stress and relaxation, methods for coping with CVD and behavioral and lifestyle change. The GCR sessions were conducted at a local university gymnasium and were performed in groups of up to 15 participants, as recommended by the German Federal Association for Rehabilitation.

Individualized combined exercise (ICE): The ICE group participated in once-weekly individualized combined resistance-endurance exercise training for 60 minutes and once-weekly traditional group-based cardiac rehabilitation as described above. The ICE intervention included 30 minutes of endurance exercise at 60-70% VO2peak and RPE 11-14 and five resistance exercises (chest press, leg press, lat pull-downs, shoulder press and seated cable row) following the recommendations of the German Federation for Cardiovascular Prevention and Rehabilitation (DGPR) and targeting the large muscle groups at an RPE<16. For the first three months, patients performed two sets of 12-25 repetitions at 30-50% 1RM; after three months patients were retested and thereafter performed two sets of 8-15 repetitions at 40-60% 1RM. The ICE sessions were located at the university sports medicine rehabilitation center and performed in groups of not more than four patients. They were instructed at a maximum 2:1 participant to therapist ratio.

ELIGIBILITY:
Inclusion Criteria:

* participation in cardiac rehabilitation
* written consent
* < 1.4 watt/kgBW exercise capacity not more than 12 weeks before study begin

Exclusion Criteria:

* >= 1.4 watt/kgBW
* contraindications to exercise participation
* hospitalized for CVD within six weeks of inclusion
* acute illness/injury (e.g. fever)
* chronic drug abuse
* inability to understand study instructions
* unwillingness to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maximal exercise capacity (watt/kgBW) | six months

SECONDARY OUTCOMES:
Change from baseline in maximal exercise capacity (watt/kgBW) | 12 months
Change from baseline in anthropometric measures | six and 12 months
  Change from baseline in waist to hip circumference ratio, body mass index, percent body fat and weight.
Change from baseline in Health Relates Quality of Life (HRQoL as measured by questionnaires) | six and 12 months
  Questionnaires used: Short From 36 (SF-36), Global Mood Scale (GMS), MacNew Heart Disease Quality of Life Instrument (MacNew)
Number of patients with adverse events (AE; documented) | six and 12 months
Change in clinical symptoms (NYHA-stage, CCS-stage, number, type and dose of medications)) | six and 12 months
Change in physical activity level (based on 7-day accelerometry) | six and 12 months
  Patients will wear accelerometers for 7 days at baseline, 6 months and 12 months, and the change in physical activity level will be calculated
Change from baseline in upper and lower body muscular strength (1RM; kg) | six and 12 months
  Upper and lower body muscular strength will be measured using a chest press and a leg extension device, respectively.
Change from baseline in anthropometric measures | six and 12 months
  Change from baseline in waist to hip circumference ratio, body mass index (BMI), percent body fat (%) and weight (kg).
Change from baseline in blood pressure (Systolic and Dystolic;mmHg) | 6 and 12 months
  24-hour blood pressure will be measured using a holter BP monitor

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Christle, M.A., Principal Investigator — Klinikum rechts der Isar
Locations (1):
- Klinikum rechts der Isar/ Technische Universitaet Muenchen, Munich, Germany